CLINICAL TRIAL: NCT07389239
Title: A Phase I/IIA Study Evaluating the Safety and Efficacy of NY-ESO-1TCR/dnTGFBRII Engineered T Cells in Combination With Decitabine in Subjects With Recurrent or Treatment Refractory Ovarian Cancer and Other Advanced Malignancies
Brief Title: A Study Evaluating the Immunotherapy Treatment for Ovarian Cancer and Other Advanced Malignancies.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1721
Record Dates: First submitted 2026-01-14; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer; Advanced Malignant Solid Tumor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Decitabine; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lead-in cohort (Experimental): Up to 6 participants will be enrolled to this arm to determine if the study treatment is safe.
  Interventions: Drug: Decitabine; Drug: Cyclophosphamide Conditioning; Biological: NY-ESO-1 TCR/ dnTGFβRII; Drug: Aldesleukin
- Dose Level -1 (Experimental): If the dose tested in Lead in cohort is not found to be safe, the dose of the NY-ESO-1 TCR/ dnTGFβRII cell dose will be lowered and up to 6 participants will be enrolled to this arm.
  Interventions: Drug: Decitabine; Drug: Cyclophosphamide Conditioning; Biological: NY-ESO-1 TCR/ dnTGFβRII; Drug: Aldesleukin
- Expansion Cohort A (Ovarian) (Experimental): Up to 6 participants with Ovarian Cancer will be enrolled to this arm after the safe dose of NY-ESO-1 TCR/ dnTGFβRII cell is found.
  Interventions: Drug: Decitabine; Drug: Cyclophosphamide Conditioning; Biological: NY-ESO-1 TCR/ dnTGFβRII; Drug: Aldesleukin
- Expansion Cohort B (Other Solid Tumors) (Experimental): Up to 6 participants with other solid tumor cancers will be enrolled to this arm after the safe dose of NY-ESO-1 TCR/ dnTGFβRII cell is found.
  Interventions: Drug: Decitabine; Drug: Cyclophosphamide Conditioning; Biological: NY-ESO-1 TCR/ dnTGFβRII; Drug: Aldesleukin

INTERVENTIONS:
Drug: Decitabine — Decitabine taken by mouth 15 mg/m2/day x 5 days, IV; Days -10 to -6
Drug: Cyclophosphamide Conditioning — Cyclophosphamide Conditioning will be 45 mg/kg x 2 days IV; Days -4 & -3
Biological: NY-ESO-1 TCR/ dnTGFβRII — The dose of NY-ESO-1 TCR/ dnTGFβRII to be tested will vary depending on assigned arm.
Drug: Aldesleukin — Aldesleukin taken by mouth500,000 IU/m2 SC BID; Days +1 to +10
  Other Names: (IL-2)

SUMMARY:
This phase I/IIA trial studies the side effects and best dose of gene-modified T cells when given with or without decitabine, and to see how well they work in treating patients with malignancies expressing cancer-testis antigens.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years and older) with histologically or cytologically of advanced (metastatic or inoperable) advanced solid tumors.
* Tumor (either an archival specimen or a fresh biopsy) shows NY-ESO-1 expression of 1+ by IHC (H-score). NY-ESO-1 expression must be confirmed by central validated assay.
* Patients with NY-ESO-1 expressing solid tumors will be included. Patients must have received, been intolerant of, or been ineligible to receive at least 2 lines of the current standard of care therapy including but not limited to chemotherapy, immunotherapy and/or targeted therapy when appropriate (e.g. Atezolizumab is approved for use in patients with alveolar soft part sarcoma) according to their disease:
* Inoperable or metastatic (advanced) ovarian, primary peritoneal or fallopian tube carcinoma:
* Has received platinum containing chemotherapy and has platinum refractory or resistant disease that has progressed on second line therapy
* If platinum sensitive disease, should have received ≥2 lines of chemotherapy.
* May have received PARP inhibitors, bevacizumab or other targeted VEGF inhibitor therapy
* Inoperable or metastatic (advanced) soft tissue sarcoma:
* Subjects must have previously received either an anthracycline or ifosfamide containing regimen.
* Gastrointestinal stromal tumors are eligible, but only must have previously received KIT-targeted therapy if a sensitizing mutation is present.
* Angiosarcomas are eligible, but only must have received prior taxane-based chemotherapy
* Urothelial carcinoma:
* Subjects must have received or refused 1 prior platinum-based therapy for the treatment of metastatic or locally advanced unresectable disease.
* Subjects who are not eligible for a platinum-containing regimen or who have progressed on a platinum-containing regimen
* Subjects may have received an anti-PD-l/PDL1 checkpoint inhibitor
* Metastatic castration-resistant adenocarcinoma of the prostate (CRPC) defined as serum testosterone level ≤ 50 ng/dL with prior surgical castration or ongoing androgen deprivation, with progressive disease:
* Progressive disease is defined by rising prostate specific antigen (PSA) or radiographic imaging according to the PCWG3 criteria during or following the direct prior line of therapy in the setting of medical or surgical castration
* At least one prior chemotherapy regimen in the metastatic setting
* Prior therapy with at least one standard 17α lyase inhibitor or second generation anti-androgen therapy for the treatment of castrate- resistant prostate cancer.
* Breast Cancer
* Prior standard of care regimens with at least one anthracycline or taxane-based regimen in either an adjuvant or metastatic setting unless intolerant or clinically not indicated. For ER positive HER2 negative cancer must have progressed on therapy with CDK 4/6 inhibitor combination. Prior hormonal therapy or Human epidermal growth factor receptor-2 (HER2) targeted therapies are allowed.
* Melanoma
* A PD-1 or PD-L1 inhibitor (with or without a cytotoxic T lymphocyte-associated protein 4 [CTLA-4] inhibitor). Patients with an actionable mutation (e.g., BRAF) must have received at least one targeted therapy.
* Non-small cell lung cancer
* A PD-1 or PD-L1 inhibitor and for patients with a PD-L1 tumor proportion score (TPS) < 50%, a platinum-based chemotherapy regimen. Patients with non-squamous NSCLC with an actionable mutation (e.g., EGFR, ALK, ROS-1) must have received at least one targeted therapy. A checkpoint inhibitor is not required for patients with actionable mutations.
* Additional advanced solid tumor expressing NY-ESO-1 are included. Patients must have received a minimum of one prior therapy.
* Subjects who are intolerant to required prior therapies must have previously received at least one systemic therapy that was deemed ineffective by the treating physician.
* At screening, must have tissue available for NY-ESO-1 testing (if not previously performed) or be willing and able to undergo a fresh tissue biopsy.
* HLA-A*0201 (HLA-A2.1) positivity by molecular subtyping (blood test or buccal swab, historical documentation acceptable).
* Age ≥ 18 years old.
* Life expectancy greater than 3 months assessed by a study physician.
* Have been informed of other treatment options.
* A minimum of one measurable lesion defined as meeting the criteria for measurable disease according RECIST1.1 criteria.
* No restriction based on prior treatments provided they have discontinued therapy at least 4 weeks prior to starting study treatment. Lesions amenable to radiotherapy or palliative radiotherapy (e.g.- bone metastases or metastases causing nerve impingement) should be treated > 4 weeks prior to enrollment and patients must be fully recovered from the effects of radiation prior to receiving the investigational agent and that patients must not receive radiation while enrolled on this study.
* Patients must have received prior anti-cancer treatment(s) or an investigational product(s) within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study treatment(s) AND unresolved or unstable serious toxic side-effects of prior chemotherapy/treatment must have recovered to Grade 1 per CTCAE (v5.0)
* Must have adequate venous access for apheresis and must be willing to and able to go through the procedure.
* Women of childbearing potential must agree to use effective methods of birth control for the duration of the study and 6 to 12 months after until persistence of the study drug is no longer detected in the peripheral blood. Methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception. It is recommended that a combination of two methods be used.
* ECOG performance status ≤1 (Karnofsky ≥80%, see Appendix A).
* Patients must have normal organ and marrow function as defined below:
* leukocytes ≥3,000/mcL
* absolute neutrophil count ≥1,000/mcL
* platelets ≥100,000/mcL
* total bilirubin ≤1.5 × ULN (institutional upper limit of normal)
* AST(SGOT)/ALT(SGPT) ≤2.5 × ULN (institutional upper limit of normal)
* creatinine ≤2 × ULN (institutional upper limit of normal) OR
* creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels > 2 × ULN
* Patient must understand the investigational nature of this study and be willing to sign a written informed consent form prior to receiving any study related procedure.
* Participant must agree to and arrange for a caregiver (age ≥ 18 years old) available 24 hours a day/ 7 days a week and arrange for lodging within 45 minutes-drive to UChicago and transportation for a period of time after discharge from the hospital. The exact amount of time will depend on the individual status as determined by the treating physician.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure with New York Heart Association class III or IV disease, patients with a LVEF < 45%, a myocardial infarction within 6 months prior to study entry or a history of myocarditis, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active autoimmune disease requiring doses of corticosteroids of ≥ 10 mg/day of prednisone (or its equivalent) or other immunosuppressive treatments.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin.
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 4 weeks prior to enrollment (inhaled or topical steroids at standard doses or isolated use of steroids as premedication for medical procedures to minimize allergic reaction [e.g. CT scan dye] are allowed).

Known cases of clinically active brain metastases (brain MRI as clinically indicated) because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment.

* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Pregnancy or breast-feeding. Patients must be surgically sterile or be postmenopausal for two years,or must agree to use effective contraception during the period of treatment and after as stated in inclusion 3.1.9. Patients with reproductive potential must have a negative pregnancy test (serum/urine) within 48 hours from starting the conditioning chemotherapy.
* Lack of availability of a patient for immunological and clinical follow-up assessment.
* Patients with pulmonary function test abnormalities as evidenced by a FEV1/FVC<70% of predicted for normality will be excluded.
* Patients with baseline O2 saturation <90% on room air.
* Patients with history of pneumonitis and/or interstitial lung disease.
* Patients with ascites, pleural or pericardial effusions which requires repeated (2 within 4 weeks) or continuous paracentesis, thoracentesis or pericardiocentesis within last 2 months.
* Patients that have had "any major surgical procedure (planned or anticipated) within 4 weeks from the first dose of study treatment(s).
* Patients who have received any live vaccines within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-06-23 (Estimated); Primary Completion 2031-12-10 (Estimated); Study Completion 2031-12-10 (Estimated)

PRIMARY OUTCOMES:
Evaluating the Safety and tolerability of autologous using immune- related Response Evaluation Criteria in Solid Tumors (irRECIST). | 2 years
  To evaluate the safety and tolerability of the autologous NY-ESO-1/ dnTGFβRII engineered T cell therapy in combination with decitabine and low-dose IL2 in patients with advanced malignancies. The irRECIST will be used for tumor response assessment performed at 6 weeks, 3 months, 6 months and 9 months.

SECONDARY OUTCOMES:
To evaluate modified cells using immune- related Response Evaluation Criteria in Solid Tumors (irRECIST). | 2 years
  To evaluate the persistence of genetically modified cells in the peripheral blood, and at tumor sites (where available). The irRECIST will be used for tumor response assessment performed at 6 weeks, 3 months, 6 months and 9 months.
Objective response rate (ORR) tumor effect | 6 weeks, 3 months, 6 months and 9 months.
  To examine the effect of the treatment on tumor as measured by objective response rate (ORR) assessed by immune- related Response Evaluation Criteria in Solid Tumors (irRECIST).
Progression free survival (PFS) tumor effect | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 9 months.
  To examine the effect of the treatment on tumor as measured by progression free survival (PFS), assessed by immune- related Response Evaluation Criteria in Solid Tumors (irRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Olson, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States